CLINICAL TRIAL: NCT07211945
Title: Loneliness as a Risk Factor for Dementia in Patients With Mild Cognitive Impairment: A Prospective Study
Brief Title: Loneliness as Risk Factor for Dementia
Acronym: SOLETE
Status: Not yet recruiting | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG-80
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Impairment (MCI); Dementia (Diagnosis); Loneliness
Keywords: Cognitive Dysfunction; Dementia; Loneliness
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Loneliness positive: Patients with mild cognitive impairment (MCI) and loneliness
- Loneliness negative: Patients with mild cognitive impairment (MCI) without loneliness

SUMMARY:
This study aims to determine whether loneliness is associated with a higher incidence of dementia in older adults with a prior diagnosis of mild cognitive impairment after 12 months of follow-up.

ELIGIBILITY:
Inclusion criteria

Patients may be included in the study if they meet all of the following criteria:

Men and women aged 70 years or older.

Diagnosis of mild cognitive impairment according to Petersen's criteria within the past 12 months.

Follow-up of the condition under study at the Alzheimer's Disease and Other Dementias Unit of Garraf (UMAG) at the Consorci Sanitari Alt Penedès-Garraf (CSAPG).

Expected follow-up of the condition at the study center.

Ability to collaborate in the required assessments.

Legal capacity to provide informed consent.

Signed informed consent for inclusion in the study, either by the participant or their legal representative.

Exclusion criteria

Participants will be excluded from the trial if they meet any of the following criteria:

Diagnosis of any of the following conditions:

Dementia: the evaluating physician will rely on the diagnostic criteria of the Spanish Society of Neurology (SEN) and the results of the neuropsychological assessment performed at the UMAG.

Participation in another study involving an experimental intervention during the present trial period and/or requiring a visit schedule incompatible with this trial.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older people affected by mild cognitive impairment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Dementia | 12 months
  Number of patients who show clinical progress from MCI to dementia

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sant Antoni Abat, Vilanova i la Geltrú, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.